CLINICAL TRIAL: NCT06113146
Title: Impact of the Eating Rate of Ultra-processed Foods on Dietary Intake Behavior and Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Next Food Collective (previously TKI agri-food program and TiFN, Top Institute Food and Nutrition) (Unknown)
Responsible Party: Principal Investigator, Ciaran Forde, prof.dr. CG (Ciarán) Forde, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RESTRUCTURE- Revamp Study
Record Dates: First submitted 2023-10-18; First posted 2023-11-02 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-06

CONDITIONS: Eating Rate
Keywords: Eating rate; Food texture; Eating behaviour; Ultra-Processed Foods; Metabolism
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The study is a balanced-order, block randomized controlled cross-over trial with 2 treatment arms. The study will have a run-in period to determine dietary habits at baseline and a washout period (14 days) to prevent carry-over effects. All participants will receive both treatments and are their own control (within participant design).
Who Masked: Participant, Outcomes Assessor
Masking Description: To cover the true aim of the study, participants will be told that the study is about different types of protein and body composition changes and that this is not a weight-loss study. Participants will be debriefed about the true study aim by email when the last participant finishes the study.
  Equal numbers of participants will be randomly allocated to each treatment order. The allocation sequence will be concealed until participants are enrolled and assigned to the intervention orders. Meals will be given a 3 random-digit code to conceal treatment allocation. However, the diets cannot be administered in a fully blinded manner due to the nature of the study foods. Study participants and research staff involved in food provision might be able to identify differences between the diets based on the types of foods served.
  Data is blinded by an independent researcher outside of the research project and unblinding will occur after the primary analyses have been conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultra-processed slow eating rate diet then the ultra-processed fast eating rate diet (Experimental): Participants assigned to this arm will receive an ultra-processed slow eating rate diet for two weeks, followed by a two week washout period and a two week ultra-processed fast eating rate diet.
  Interventions: Other: ultra-processed slow eating rate diet; Other: Ultra-processed fast eating rate diet
- ultra-processed fast eating rate diet then the ultra-processed slow eating rate diet (Experimental): Participants assigned to this arm will receive an ultra-processed fast eating rate diet for two weeks, followed by a two week washout period and a two week ultra-processed slow eating rate diet.
  Interventions: Other: ultra-processed slow eating rate diet; Other: Ultra-processed fast eating rate diet

INTERVENTIONS:
Other: ultra-processed slow eating rate diet — Consuming ultra-processed slow eating rate meals (served ad libitum) and snacks. Eating rate is manipulated through food texture, for example foods with a hard texture that require a long chewing duration before a bite of food can be swallowed.
Other: Ultra-processed fast eating rate diet — Consuming ultra-processed fast eating rate meals (served ad libitum) and snacks. Eating rate is manipulated through food texture, for example foods with a soft texture that require little chewing before a bite of food can be swallowed.

SUMMARY:
The aim of this balanced-order block randomized controlled cross-over trial with 2 treatment arms is to determine the effect of eating rate (ER) of ultra-processed food diets (UPF fast ER vs UPF slow ER) on ad libitum energy intake across a two week period.

DETAILED DESCRIPTION:
Rationale: Consumption of industrially processed foods has been associated with obesity and related adverse health outcomes. If this reflects a causal relationship, it is unknown what attributes or properties of industrially processed foods might drive this association. Extensive research has shown that foods consumed with a texture-derived slow eating rate (ER) are consumed in smaller amounts relative to foods consumed with a fast ER. ER has been suggested as one of the mechanisms why (ultra-)processed foods (with a fast ER) may promote excess in calorie intakes. We will therefore test the hypothesis that ER moderates energy intakes from ultra-processed foods.

Objective: The primary objective of this study is to determine the effect of ER of ultra-processed food diets (UPF slow ER vs UPF fast ER) on ad libitum energy intake (kcal/day) across a two week period. The secondary objectives are to compare body composition and metabolic changes that occur when on a 14 day diet of ultra-processed foods with either a slow or a fast ER.

Study design: We will conduct a balanced-order, block randomized controlled cross-over trial with 2 treatment arms, to determine the effect of ER of ultra-processed food diets (UPF fast ER vs UPF slow ER) on ad libitum energy intake (kcal) across a two week period. The study will have a run-in period to determine habitual dietary habits (baseline) and a washout period (14 days) between treatments to prevent carry-over effects. All participants will receive both treatments and are their own control (within subject design).

Study population: 39 healthy, non-smoking, adults between 21-50 years old and with a BMI between 21-27 kg/m2 will be included.

Intervention: The two treatments are 1) a 14-days ultra-processed, slow ER diet, and 2) a 14-days ultra-processed, fast ER diet. The ad libitum meal menus are matched for energy density (kcal/g), liking (hedonic range), and level of processing, but different in textural characteristics known to influence ER. During the treatment periods participants eat all of their main meals at the research site on weekdays. Participants receive pre-packed meals to consume at home for the weekends. Meals are served ad-libitum, presented in portions that are > 200% of a regular portion size. Participants are asked to eat from each meal until they feel comfortably full. Food (gram) and energy (kcal) consumed will be recorded at the level of the meal, the day and week of the interventions.

Main study parameters/endpoints: The primary outcome is the between-treatment difference in average (across 14 days) daily energy intake (kcal/day). Secondary study parameters include between-treatment differences in: food intake (g/day), body weight and body composition changes, postprandial hormone responses and respiratory quotient changes to a mixed meal tolerance test, continuous measures of glucose levels, and changes in fasted state leptin and ghrelin levels and blood lipid profiles.

ELIGIBILITY:
In order to be eligible to participate in this study, a participant must meet all of the following criteria:

* Between 21-50 years old at the day of inclusion
* Being able to read and understand English
* BMI 21-27 kg/m2
* Good general and mental health and appetite (self-report)
* Commonly (5 out of 7 week days) eating three meals a day around approximately the same times (self-report).

A potential participant who meets any of the following criteria will be excluded from participation in this study:

Based on the information meeting:

* Difficulties with swallowing, chewing and/or eating in general
* Suffering from an endocrine or eating disorder, gastrointestinal illness or illness of the thyroid gland, cardio-vascular diseases, bowel diseases, respiratory disease, neurological diseases, or diabetes, anaemia, cancer, or psychiatric conditions such as clinical depression, burnout or anxiety or bipolar disorder.
* Having a history of low blood pressure
* Having taste or smell disorders (self-report)
* Braces (not including a dental wire) or oral piercing
* Followed an energy restricted diet during the last 2 months
* Currently using or in the past 3 months (calculated from the first day of the study) used prebiotics supplements, probiotic supplements and/or antibiotics
* Gained or lost 5 kg of body weight over the last half year
* High restrained eater (DEBQ restrained eater scale ≥ 2.90 for males and ≥ 3.40 for females [23])*
* Use of medication, including but not limited to hormone therapy or medications that affect the immune system or any medication that influences study outcomes such as food intake, appetite in general or metabolic responses (self-report)
* Consuming on average more than 21 (men) or 14 (women) glasses of alcohol per week
* Pregnant or lactating women, or women who are planning on becoming pregnant within the study period.
* Smoking (daily)
* Not willing to stop using drugs during the study period (from inclusion till last test session)
* Not willing to stop consuming alcohol during the intervention weeks
* Exercising more than 4 hours per week (excluding biking and walking at a normal pace and distance)
* Following a vegetarian or vegan diet
* Allergies or intolerance to any ingredient of the test meals
* Not willing to eat the test food because of eating habits or believes
* Do not like > 20% of the test foods or its ingredients based on descriptions of the meal (scoring items ≤ dislike on a nine point hedonic scale)*
* Majority > 50% of dietary food intake (g) is derived from ultra-processed foods (based on a food frequency questionnaire (FFQ) based on normative data collected in pre-trial.* The 50% cut-off is based on median intake of UPFs in Dutch cohort studies [24] [25]
* Being unfamiliar with > 25% of the test meals
* Signed up for participating in another research study
* Being an employee or thesis student of the Division of Human Nutrition and Health at Wageningen university
* Radiological investigation during past 7 days where iodine or barium containing contrast fluids have been used (DEXA contra-indication)
* Nuclear medical investigation involving isotopes during past 7 days (DEXA contra-indication)

Exclusion after screening:

* Haemoglobin value is not between 7.5-11.0 mmol/L (women), 8.5-11.0 mmol/L (men)
* Fasted glucose level is below < 3.5 mmol/L or higher than 8 mmol/L
* Blood pressure is below 90/60 mm hg (below 90 and/or below 60 mm hg)
* Veins are not suited for blood sampling (as judged by trained research nurses)
* Persons with an extremely fast or slow eating rate trait, (> 2 times the SD from the median, based on the carrot test [26] eating rate distribution based on data collected in previous studies in the same study population (unpublished).
* Persons with little difference (< 20%) in the eating rate of a hard or soft carrot
* Do not like > 20% of the test foods based tasting small portions (1 bite) of each of the meals (scoring items below ≤ dislike on a nine point hedonic scale)* * This exclusion criterion will not explicitly be communicated to the participants to prevent desirable answers

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Average daily energy intake (kcal/day) | Two periods of 14 days
  The average (across two weeks) daily energy intake (kcal/day) in each diet arm

SECONDARY OUTCOMES:
Total Energy intake (kcal) | Two periods of 14 days
  Ad libitum energy intake (kcal) per meal, day and week.
Total Food intake (gram) | Two periods of 14 days
  Ad libitum food intake (gram) per meal, day, week and average daily food intake (gram/day) in each diet arm.
Cumulative energy intake (kcal) | Two periods of 14 days
  Cumulative energy intake (kcal) over the study period (14 days)
Cumulative food intake (gram) | Two periods of 14 days
  Cumulative food intake (gram) over the study period (14 days)
Body weight (kg) | Pre and post intervention periods and six times (every other day) during each intervention period of 14 days
  Participant's weight will be measured in duplicate to obtain an average. The participant will be measured in stocking feet and light clothing on a standard balance scale. Participant will not be able to see their weight.
Total and Regional Fat Mass and Fat Free Mass (kg, %) | Pre and post 14-day intervention periods
  Changes in fat mass and fat free mass (kg, %) will be measured using; DEXA, air displacement plethysmography (BODPOD), skinfold measurements
Postprandial hormone responses (Mixed Meal Tolerance Test) | Baseline and post 14-day intervention periods
  Insulin and glucose, total ghrelin, total GLP-1, PP, PYY, Glucagon and c-peptide responses, to a fixed calorie test meal (rice porridge)
Metabolic outcomes (Mixed Meal Tolerance Test) | Baseline and post 14-day intervention periods
  Resting energy expenditure will be measured 30 minutes before a Mixed Meal Tolerance Test (MMTT) consisting of a fixed energy amount of rice porridge, and 30 minutes immediately after the meal using a ventilated hood. Based on this we will estimate the respiratory quotient, diet induced thermogenesis and substrate use. Based on the resting energy expenditure in combination with physical activity levels (estimated based on accelerometer (actigraphy) and 24hr recalls of exercise/sports) energy expenditure will be calculated per participant.
Glucose Excursions | Every 15 minutes throughout two 14-day intervention periods
  24-hour glucose levels will be measured using Continuous Glucose Monitoring (CGM). This will be used for a comparison of percentage of time spent within and out of the normative range.
Leptin and Ghrelin levels (Fasted state) | Baseline and post 14-day intervention periods
  Leptin, Ghrelin blood plasma concentrations after an overnight fast
Blood lipid profile (Fasted state) | Baseline and post 14-day intervention periods
  Total cholesterol, HDL, LDL, free fatty acids and other blood lipids

OTHER OUTCOMES:
Eating behaviour observed during meals of intervention diets using video-annotation | Two periods of 14 days
  Total meal duration (min), bite duration (min) and number of bites
Derived measures of eating behaviour observed during meals of intervention diets using video-annotation | Two periods of 14 days
  Derived measures of eating behaviour such as eating rate (g/min) based on video-annotation.
Micro-structure of eating observed during meals of intervention diets using video-annotation | Two periods of 14 days
  Chewing behaviour, oro-sensory exposure time, bite size (gram/bite) and bite frequency (bite/min) based on video-annotation.
Eating behaviour observed during meals of intervention diets using weighing tray | Two periods of 14 days
  Eating behaviour characteristics (eating rate (gram/min), total meal duration (min), bite duration (min), bite frequency (bite/min), number of bites (per meal), bite size (gram/bite), oro-sensory exposure time (seconds/bite), cumulative weight change of the meal from start to end, based on weighing tray.
Sensory attributes of intervention meals | pre and post meals during two 14-day intervention periods
  Sensory properties, liking and familiarity of the meals, assessed after one bite of each meal on a 100mm Visual Analogue Scale ranging from "Not at all" (0mm) to "Extremely" (100mm).
Macro-nutrient intake (grams and %EN) | Two periods of 14 days
  Intake of carbohydrates, protein, and fat (gram; %EN) per meal, day, week and study period.
Dietary intake during washout periods | At baseline and washout; 3 days
  Dietary intake (energy intake, macronutrients, fiber, salt, and UPF) will be measured using a 3 day food diary ( 2 week-days and one weekend day).
Sodium and nitrogen in urine (24 hr urine sample collection) | 4 x 24 hours during the intervention periods and 4 times urine sample collection during the two 14 day intervention periods
  Sodium and nitrogen in urine will be measured in urine as markers for salt and protein intake as compliance markers of participants dietary intakes
Urine metabolites (24 hr urine sample collection) | 3x24hr urine collection once at baseline and post both 14-day intervention periods
  Untargeted metabolomics, C-peptide, creatinine
Nutrient intake (grams and %en) during intervention periods | Two periods of 14 days
  Intake of mono- and disaccharides, fibre (grams, gram/100 kcal) and salt (grams, gram/100kcal) per meal, day, week and study period
Dutch Healthy Diet index 2015 | At baseline, two periods of 14 days and washout
  Dutch Healthy Diet index 2015 (DHD15-index) consists of fifteen components each representing one of the fifteen food-based Dutch dietary guidelines (2015). Per component the score ranges from 0 to 10, resulting in a final total range score between 0 (no adherence) and 150 (complete adherence).
Subjective appetite | pre and post meals during two 14-day intervention periods
  Summary of questions on participants' perceived level of hunger, fullness, thirst and the desire to eat indicated on 100mm Visual Analogue Scales ranging from "Not at all" (0mm) to "Extremely" (100mm).
Adiposity distribution | Pre and post 14-day intervention periods
  Waist to hip ratio circumference will be calculated by dividing the waist measurement (cm) by the hip measurement (cm).
Water retention | Pre and post 14-day intervention periods
  Changes in water retention (kg, %) will be measured using bio impedance analysis (BIA)
Glucose level (various outcomes) | Two periods of 14 days
  24-hour glucose levels will be measured every 15 minutes using Continues Glucose Monitoring (CGM).
HbA1c | Baseline; 10 minutes
  Blood HbA1c
Resting energy expenditure | Baseline and post 14-day intervention periods
  VO2 and VCO2 measures will be measured using the ventilated hood for 30 minutes
Person trait: oral processing behaviour | Screening; 5 minutes
  Standardized method to determine oral processing behaviour as a personal trait (Carrot test).
Appetitive Traits (study population characteristics): Dutch Eating Behaviour Questionnaire | Screening; 15 minutes
  The Dutch Eating Behavior Questionnaire (DEBQ) consists out of 33 questions which can be scored from "Never" (1) to "Very often" (5) and will be used to classify participants based on their eating behavior trait (restrained eater, emotional eater, external eater). High restrained eaters will be identified with DEBQ restrained eater scale ≥ 2.90 for males and ≥ 3.40 for females.
Appetitive Traits (study population characteristics): Adult Eating behaviour questionnaire | Screening; 15 minutes
  The Adult Eating Behaviour Questionnaire (AEBQ) will be used to characterize the appetitive traits of the participants. The questionnaire consists out of 35 statements which can be scored from "Strongly agree" (1) to "Strongly disagree" (5). The statements are summarized into the scales 'Enjoyment of food', 'Emotional over-eating', 'emotional under-eating', 'Food fussiness', 'Food responsiveness', 'Hunger', 'Slowness in eating', and 'Satiety responsiveness'.
Appetitive Traits (study population characteristics): Reasons Individuals Stop Eating Questionnaire | Screening; 5 minutes
  The Reasons Individuals Stop Eating Questionnaire (RISE-Q15) consists out of 15 questions in which the reasons or eating cessation can be assessed. All items are scored on a 7-point frequency scale (Never, Rarely, Seldom, Sometimes, Often, Usually, and Always) and summarized into 5 subscales: decreased food appeal, physical satisfaction, planned amount, self-consciousness, and decreased priority of eating.
Person trait: Interoceptive awareness | Screening; 15 minutes
  The conscious level of interception with its multiple dimensions potentially accessible to self-report will be accessed with the Multidimensional Assessment of Interoceptive Awareness version 2 (MAIA-2). MAIA-2 is a validated 8-scale state-trait questionnaire with 37 statements. The statements are scored from "Never" (0) to "Always" (5). The scales are 'Noticing', 'Not-Distracting', 'Not-Worrying', 'Attention regulation', 'Emotional Awareness', 'Self-Regulation', 'Body Listening', and 'Trusting'.
Diet Satisfaction | Baseline and post 14-day intervention periods
  The satisfaction of the participants with the diets (baseline, UPF fast and UPF slow) will be assessed with the Diet Satisfaction Questionnaire (Dsat-28) [40]. The Dsat-28 is a validated questionnaire that consists out of five scales accessed by 28 statements about the characteristics of the lifestyle and attitudes of individuals that reflect satisfaction within the diets. The agreement to the statements will be scored from "Disagree strongly" (1) to "Agree strongly" (5). The scales are 'Healthy Lifestyle', 'Eating Out', 'Costs', 'Preoccupation with Food', and 'Planning and preparation' . Only questions that are applicable will be asked (e.g. for the test diets no questions belonging to the scales Costs or Eating Out will be asked).
Habitual dietary intake at baseline | At baseline covering past 14 days
  Using the Food Frequency Questionnaire (FFQ) the dietary intake at baseline will be measured in terms of macro(nutrients) and NOVA class.
Person trait: Salivary flow | Baseline; 15 minutes
  Alpha-amylase activity and stimulated saliva flow rate
Blood pressure (fasted state) | Baseline and post 14-day intervention periods
  measured in mm/hg after an overnight fast
Physical activity: accelerometry | Two periods of 14 days
  Physical activity will be measured using accelerometry
Physical activity: exercise diary | Two periods of 14 days
  Physical activity will be measured using exercise diaries
Physical activity questionnaire | Baseline; 10 minutes
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) records the activity of the last 7 days on four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. It estimates energy expenditure based on reported physical activity.
Markers of gut health | Baseline and post 14-day intervention periods
  Inflammatory and leaky gut markers will be measured by measuring changes in C-reactive protein (CRP), IL-6, IL-8, TNF-α,levels of zonulin, gamma-glutamyltransferase, leukocytes, lipopolysaccharide-binding protein, soluble CD14, bactericidal increasing protein, peptidoglycan in fasted state.
Bolus properties (person characteristic) | Baseline and post 14-day intervention periods
  The bolus properties the mixed meal tolerance test will be analysed on total number, surface area (mm2), and particle size (mm2 or mm).
Bolus saliva uptake (person characteristic) | Baseline and post 14-day intervention periods
  The bolus properties the mixed meal tolerance test will be analysed on the amount of saliva uptake (g).
Microbiome | Pre and post 14-day intervention periods
  Measuring of fecal metabolite profile (SCFAs, tryptophan metabolites and bile acids), metagenomics, microbiota composition, and water content of fecal samples
Gut transit time | Pre and post 14-day intervention periods
  Measure of gut transit time using the blue dye test
Gastrointestinal symptoms | Baseline and post 14-day intervention periods
  The Irritable bowel syndrome severity scoring system (IBS-SSS) will be used to assess the severity of IBS (gastrointestinal symptoms). The IBS-SSS consists of five questions in which severity of IBS symptoms in the last 10 days will be assessed on a 0 - 100 VAS scale. The sum of the scores of these five questions indicate the severity of IBS with a maximum achievable score of 500. Scores of 75 - 175 indicate a mild form of the disease, 175-300 a moderate form and scores of 175-300 indicate a severe type of IBS.
Stoolform | Baseline and post 14-day interventions periods
  Participants will be asked classify their stool on the Bristol Stool Form Scale (BSFS). The BSFS is a 7-pont scale. The BSFS is an ordinal scale of stool types ranging from the hardest (Type 1) to the softest (Type 7). Types 1 and 2 are considered to be abnormally hard stools while Types 6 and 7 are considered abnormally loose/liquid stools. Type 3, 4 and 5 are therefore generally considered to be the most 'normal' stool form and are the modal stool forms in cross-sectional surveys of healthy adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available according to the FAIR principles on Open Science Framework (OSF)
Supporting Information: SAP, Analytic Code
Time Frame: Prior to data analyses
Access Criteria: Statistical Analysis Plan and the Analytic Code will be made available at OSF
URL: https://osf.io/afmkh

REFERENCES:
- [Derived] Forde CG, Heuven LA, van Bruinessen M, Liu Z, Stieger M, de Graaf K, Lasschuijt MP. Eating rate has sustained effects on energy intake from ultraprocessed diets: a 2-week ad libitum dietary randomized controlled crossover trial. Am J Clin Nutr. 2025 Nov 26:101122. doi: 10.1016/j.ajcnut.2025.11.012. Online ahead of print. PMID 41314613
- [Derived] Lasschuijt MP, Heuven LAJ, van Bruinessen M, Liu Z, Rubert J, Stieger M, de Graaf K, Forde CG. The Effect of Eating Rate of Ultra-Processed Foods on Dietary Intake, Eating Behaviour, Body Composition and Metabolic Responses-Rationale, Design and Outcomes of the Restructure Randomised Controlled Trial. Nutr Bull. 2025 Dec;50(4):640-655. doi: 10.1111/nbu.70027. Epub 2025 Sep 9. PMID 40926558
- See also: Project webpage — https://restructureproject.org/